CLINICAL TRIAL: NCT04718246
Title: Stability Of Dental Implants Placed In Healed Bony Sites Of Hyperlipidemic Patients: A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maie Ismaiel mohammed Fathy, Assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Maie2
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Implant Stability
Keywords: Hyperlipidemia; Implant survival; osseointegration; CBCT
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental Implants in hyperlipidemia patients (Other): Implants will be placed at T0, then Implant site exposure will take place 6 months following the implant placement. Insertion of the healing collars in order to obtain adequate soft tissue form for 1-2 weeks then the impressions (indirect, closed tray echnique) shall be taken to fabricate the final crowns, then the final crowns will be fitted in place.
  Interventions: Other: Dental Implants Placed In hyperlipidemia patients

INTERVENTIONS:
Other: Dental Implants Placed In hyperlipidemia patients — A preoperative cone beam CT (CBCT) will be performed for each patient prior to the surgery.
  Surgical phase (T0):
  After local anesthetics, all osteotomies will be prepared by the same operator, using a drilling speed of 1200 rpm, under copious irrigation with normal saline.
  * Penetration of cortical bone will be achieved with no. 6 round burs.
  * The osteotomies will be widened, using a drill 1 mm larger than the final drill provided by the manufacturer. The final size of the control osteotomies were same diameter of the implant.
  * Periotest® will measure initial implant stability. Implant site exposure will take place 6 months following the implant placement. Insertion of the healing collars in order to obtain adequate soft tissue form for 1-2 weeks

SUMMARY:
Statement of the problem:

Osseo-integration of dental implants depends mainly on bone regeneration around dental implant. Hyperlipidemia has significant adverse effects on bone health, leading to lower bone mineral density and to higher risk of osteoporosis and bone fracture (Corwin 2003; Pirih, Lu et al. 2012). The effects of hyperlipidemia on bone health may also interfere with dental implant therapy since the host's bone quantity, quality and healing potential play an important role in osseointegration (Fedele, Sabbah et al. 2011; Gaetti-Jardim, Santiago-Junior et al. 2011; Olivares-Navarrete, Raines et al. 2012).

Rationale for conducting the research:

Hyperlipidemia has been associated with the pathophysiology of major diseases, such as atherosclerosis and osteoporosis.

A high cholesterol level has significant adverse effects on bone, including lower bone density, volume and strength. Statins, drugs that lower serum cholesterol levels have beneficial effects on bone metabolism. Since host's bone quantity, quality and healing potential play a crucial role in osseointegration of dental implants, it was hypothesized that hyperlipidemia may negatively affect implant osseointegration.

DETAILED DESCRIPTION:
The high predictability of dental implants has led to routine use with a great expectation for success. There are many researches focused on the outcome of delayed dental implant. Since the first report of highly success rate after placement of a dental implant, there has been increasing interest in this technique for implant treatment (Chen ST., 2004) The goal of modern dentistry is to restore the patient's dentition to normal contour, function, comfort, esthetics, speech and health regardless of the atrophy, disease or injury of the stomatognathic system, as a result of disease related tooth loss and the value placed upon teeth, there has been a continual search for methods by which missing teeth could be replaced. Early artificial replacements were made from natural teeth and a variety of substitute materials. All transplantation of a tooth from one person to another was an early method by which lost teeth were replaced. Archeological discoveries indicate that many ancient civilizations practiced allogenic tooth transplantation. In 1561, Ambrose Pare reported that decayed teeth could be replaced by using extracted teeth from another individual and is credited with being the first to mention transplantation (Chiu YW., 2015) Periimplant osteogenesis consists of postsurgical reaction and remodeling of the bone and the initiation and progression of de novo bone formation, which are represented as a reduction in primary stability and development of secondary stability, respectively (Ogawa and Nishimura, 2003, Aparicio et al., 2006, Atsumi et al., 2007). Dental implant survival is mainly dependent on successful osseointegration following placement. Any alteration of this biological process may adversely affect the success rate. Also, the long-term prognosis is adversely affected by inadequate bone volume at implant sites. There are several risk factors that were defined as implant failure. One of the risks of implant's failure depends on the systemic health of the subject (such as diabetes mellitus, osteoporosis, smoking) Recently, some authors suggested that there is a relationship between hypercholesterolemia and dental implant osseointegration (Keuroghlian A et al.. 2015, Tirone F et al. 2016). Hyperlipidemia is a state with an abnormal lipid pro- file, which is characterized by elevated blood concentrations of triglycerides, elevated levels of total cholesterol and LDL, and decreased levels of HDL cholesterol ( Saxlin T., 2008) Hyperlipidemia is associated with several diseases such as atherosclerosis and osteoporosis. The National Health and Nutrition Examination Survey (NHANES III) reported that 63% of osteoporotic patients have hyperlipidemia (Bilezikian JP., 2005) The main mechanisms of the relationship between hyperlipidemia and bone tissue metabolism are the involved aspects of some metabolic changes, including lower bone mineral density, increase in the number of osteoclasts, and the inhibition of osteoblastic activity. However, several investigators suggested that lipid- lowering drugs, such as statins, had beneficial effects on bone metabolism and also favorable effects on statins observed on osteogenesis around implants (Moriyama Y et al., 2010). Recently many papers focused on High cholesterol and its impact effect on bone turn over around dental implant but all of them are animal studies. Mish (2008) defined four bone density groups (D1 to D4) found in all jaw regions varying according to macroscopic cortical and trabecular bone types. D1 is dense and homogenous type of bone that is often found in anterior mandibles. D2 is a combination of dense-to-porous cortical bone on the crest and coarse trabecular bone on the inside. D3 is composed of thinner porous cortical bone on the crest and fine trabecule. Mish (2008) defined four bone density groups (D1 to D4) found in all jaw regions varying according to macroscopic cortical and trabecular bone types. D1 is dense and homogenous type of bone that is often found in anterior mandibles. D2 is a combination of dense-to-porous cortical bone on the crest and coarse trabecular bone on the inside. D3 is composed of thinner porous cortical bone on the crest and fine trabecular bone within the ridge. The D2 bone trabeculae are 40% to 60% stronger than D3 trabeculae. D4 bone has very little density and little or no cortical crestal bone. It is the opposite of D1. The most common locations for D4 type of bone are the posterior region of the maxilla. D4 bone trabeculae may be up to 10 times weaker than the cortical bone of D1 and the bone-implant contact after initial loading is often less than 25%. Bone trabeculae are sparse and, as a result, initial fixation of any implant design presents a surgical challenge (Dvorak G., 2011) Primary or secondary implant stability usually measured by Periotest or Ostell, Periotest measuring procedure is electromechanical. An electrically driven and electronically monitored tapping head percusses the implant 16 times. The entire measuring procedure requires approx. 4 seconds. The tapping head is pressure sensitive and records the duration of contact with the test object. Loose implants display a longer contact time and the Periotest values are correspondingly higher, while osseointegrated implants have a short contact time and result in low Periotest values. Periotest values (PTV) of (-8 to +50) were -ve values considered the ideal values that denote successful osseointegration (Molly L., 2006). Although the ever-increasing number of published animal studies on this topic, there is however no consensus regarding dental implants stability in patients with hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

Patients who have at least one missing tooth.

* Patient with hyperlipidemia (LDL < 160 mg/dl )
* Patients with sufficient interarch space.
* Patients aged from 20 to 60 years old.
* Good oral hygiene.(Wiesner et al. 2010)
* Accepts 6 months follow-up period (cooperative patients)
* Patient provides an informed consent.

Exclusion Criteria:

Patients with signs of acute infection related to the area of interest.

* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits (Lobbezoo et al. 2006).
* Current and former smokers (Lambert et al, 2000)
* Pregnant women.
* Psychological problems -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability | At time of implant placement, 6 months post-implant placement
  Outcome will be determined using sonance frequency analysis (RFA) (Osstell) periotest

SECONDARY OUTCOMES:
Pain | Measured 7 and 14 days post-implant placement
  Measured using Numerical Rating Scale
Swelling | 7 days post-implant placement
  Measured using verbal rating scale, categorized as either (VRS) Absent-slight-moderate- Or intense
Crestal bone level | Same day as implant placement, 3 and 6 months post-implant.
  Digital periapical radiograph using a radiographic holder and an acrylic radiographic stent -which is constructed previously on patient's cast= will be taken to determine the crestal bone level and resorption. The parallel technique in combination with the acrylic stent is performed to ensure reproducibility.
Osseointegration | Same day as implant placement, 3 and 6 months post-implant.
  Digital periapical radiograph using a radiographic holder and an acrylic radiographic stent -which is constructed previously on patient's cast= will be taken to determine the crestal bone level and resorption. The parallel technique in combination with the acrylic stent is performed to ensure reproducibility.
Implant survival | 6 months post-implant placement
  Assessed as a dicotomous outcome (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No